CLINICAL TRIAL: NCT01622790
Title: An Evaluation of the Bioequivalence of a Combined Formulated Tablet (50mg/600mg/300mg Dolutegravir/Abacavir/Lamivudine) Compared to One Dolutegravir 50mg Tablet and One EPZICOM† (600mg/300mg Abacavir/Lamivudine) Tablet Administered Concurrently and the Effect of Food on Bioavailability of the Combined Formulation in Healthy Adult Subjects
Brief Title: Evaluation of the Bioequivalence of a Combined Formulated Tablet
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: Shionogi (Industry); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 114580
Record Dates: First submitted 2012-05-31; First posted 2012-06-19 (Estimated); Last update posted 2012-10-15 (Estimated); Status verified 2012-10

CONDITIONS: Infection, Human Immunodeficiency Virus
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome | interventions — dolutegravir; abacavir; Lamivudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): 33 subjects will receive a single dose of each of a tablet formulation of dolutegravir 50 mg/abacavir 600 mg/lamivudine 300 mg in Period 1followed by dolutegravir 50 mg plus EPZICOM (abacavir 600mg/lamivudine 300 mg) in Period 2. Approximately 6 of these subjects will return for a third period where they will receive a single dose of dolutegravir 50 mg/abacavir 600 mg/lamivudine 300 mg after a high fat breakfast. There will be a screening visit within 30 days prior to first dose and a follow-up visit 7-14 days after the last dose.
  Interventions: Drug: Dolutegravir 50 mg/abacavir 600 mg/lamivudine 300 mg; Drug: Dolutegravir 50 mg; Drug: abacavir 600 mg/lamivudine 300 mg
- Arm 2 (Experimental): 33 subjects will receive dolutegravir 50 mg plus EPZICOM (abacavir 600mg/lamivudine 300 mg) in Period 1 followed by a single dose of a tablet formulation of dolutegravir 50 mg/abacavir 600 mg/lamivudine 300 mg in Period 2. Approximately 6 of these subjects will return for a third period where they will receive a single dose of dolutegravir 50 mg/abacavir 600 mg/lamivudine 300 mg after a high fat breakfast. There will be a screening visit within 30 days prior to first dose and a follow-up visit 7-14 days after the last dose.
  Interventions: Drug: Dolutegravir 50 mg/abacavir 600 mg/lamivudine 300 mg; Drug: Dolutegravir 50 mg; Drug: abacavir 600 mg/lamivudine 300 mg

INTERVENTIONS:
Drug: Dolutegravir 50 mg/abacavir 600 mg/lamivudine 300 mg — Dolutegravir 50 mg/abacavir 600 mg/lamivudine 300 mg is an experimental fixed dose combination tablet of an experimental integrase inhibitor (dolutegravir) and two FDA approved nucleoside reverse transcriptase inhibitors (abacavir and lamivudine)
Drug: Dolutegravir 50 mg — Dolutegravir is an experimental drug in the integrase inhibitor class that is being studied for the treatment of HIV infection.
Drug: abacavir 600 mg/lamivudine 300 mg — This is an FDA approved fixed dose combination tablet of two nucleoside reverse transcriptase inhibitors
  Other Names: KIVEXA. This is a trademark of ViiV Healthcare; EPZICOM. This is a trademark of ViiV Healthcare.

SUMMARY:
Dolutegravir (DTG, GSK1349572) is a next-generation integrase inhibitor (INI) currently in phase 3 clinical trials for human immunodeficiency virus (HIV). Fixed-dose combinations (FDCs) have greatly simplified the treatment of patients with HIV. While Atripla (an FDC of tenofovir (TDF), emtricitabine (FTC) and efavirenz (EFV)) has become the preferred first line regimen due in large part to its convenient presentation as a full treatment regimen in a single product, other options are needed. A fixed-dose combination of DTG/abacavir (ABC)/lamivudine (3TC) is one such opportunity. Part A of this study will be a single-dose, two-treatment crossover pivotal bioequivalence (BE) evaluation of the DTG/ABC/3TC FDC tablet in 66 healthy subjects. The reference formulations in this trial will be the 50 mg DTG tablet that is currently being used in the Phase 3 clinical trials and the already marketed FDC tablet product EPZICOM™ (ABC 600 mg/3TC 300 mg).It is intended that the results of this pivotal bioequivalence study will show that the proposed commercial DTG/ABC/3TC FDC tablet formulation is bioequivalent to DTG plus EPZICOM administered as separate tablets. Part B of this study will evaluate the effect of a high fat meal on the FDC tablet in 12 healthy subjects that have already participated in Part A of the study. There will be a screening visit within 30 days prior to the first dose of study drug and a follow up visit within 7-14 days after the last dose. There will be a 7 day washout between doses in each treatment period. The following PK parameters for DTG, ABC and 3TC will be measured: area under the concentration curve from time zero (pre-dose) extrapolated to infinite time (AUC(0-infinity)), Area under the concentration-time curve from time zero (pre-dose) to the time of the last quantifiable concentration (AUC (0-t)), maximum observed concentration (Cmax), lag time before observation of drug concentrations (tlag), time of occurrence of Cmax (tmax), terminal phase half-life (t½), terminal elimination phase rate constant (λz), percentage of AUC obtained by extrapolation (%AUCex),apparent clearance following oral dosing (CL/F) and apparent terminal phase volume

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac evaluation.
* Male or female between 18 and 55 years of age inclusive, at the time of signing the informed consent.
* A female subject is eligible to participate if she is of: Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation, bilateral salpingo-oophorectomy or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) greater than 40 mIUml and estradiol less than 40 pg/ml (less than 146.8 pmol/L) is confirmatory]. Child-bearing potential and agrees to use one of the contraception methods listed in the protocol for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until the follow-up visit.
* Male subjects with female partners of child-bearing potential must agree to use one of the contraception methods listed in the protocol. This criterion must be followed from the time of the first dose of study medication until 84 days after the last dose of study drug.
* Body weight greater than and equal to 50 kg for males and greater than and equal to 45 kg for females and BMI within the range 18.5- 31.0 kg/m2 (inclusive).
* ALT, alkaline phosphatase and bilirubin less than and equal to 1.5xULN (isolated bilirubin greater than 1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%). A single repeat is allowed for eligibility determination.
* A negative HLA-B*5701 allele screening assessment
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form

Exclusion criteria:

* The subject has a positive pre-study drug/alcohol screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* History of sensitivity to any of the study medications, or components thereof, or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety. If heparin is used during PK sampling, subjects with a history of sensitivity to heparin or heparin-induced thrombocytopenia should not be enrolled.
* History of regular alcohol consumption within 6 months of the study defined as: An average weekly intake of greater than 14 drinks/week for men or greater than 7 drinks/week for women. One drink is equivalent to (12 g alcohol) = 5 ounces (150 ml) of wine or 12 ounces (360 ml) of beer or 1.5 ounces (45 ml) of 80 proof distilled spirits.
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice from 7 days prior to the first dose of study medication.
* Pregnant females as determined by positive serum or urine human chorionic gonadotrophin (hCG) test at screening or prior to dosing.
* Lactating females.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subjects with a pre-existing condition interfering with normal gastrointestinal anatomy or motility, hepatic and/or renal function, that could interfere with the absorption, metabolism, and/or excretion of the study drugs. Subjects with a history of cholecystectomy, peptic ulceration, inflammatory bowel disease or pancreatitis should be excluded.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* A positive test for HIV antibody.
* History of Gilbert's disease.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* The subject's systolic blood pressure is outside the range of 90-140mmHg, or diastolic blood pressure is outside the range of 45-90mmHg or heart rate is outside the range of 50-100bpm for female subjects or 45-100 bpm for male subjects. A single repeat is allowed for eligibility determination.
* Exclusion criteria for screening ECG (a single repeat is allowed for eligibility determination): Heart rate: Males less than 45 and greater than 110 bpm; Females less than 50 and greater than100 bpm; PR Interval: Males less than 120 and greater than 220 msec; QRS duration: Males less than 70 and greater than 120 msec; QTc interval (Bazett): Males greater than 450 msec; Evidence of previous myocardial infarction (does not include ST segment changes associated with repolarization); Any conduction abnormality (including but not specific to left or right complete bundle branch block, AV block [2nd degree or higher], Wolf Parkinson White [WPW] syndrome), non-sustained or sustained ventricular tachycardia (greater than and equal to 3 consecutive ventricular ectopic beats), and sinus pauses greater than 3 seconds; Any significant arrhythmia which, in the opinion of the principal investigator and GSK medical monitor, will interfere with the safety for the individual subject

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2012-06; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Plasma DTG(dolutegravir), ABC (Abacavir) and 3TC(Lamivudine) PK(Pharmacokinetic) parameters, Area under the concentration-time curve from time zero (pre-dose) | For 48 hours after dosing on Day 1 of Periods 1, 2 and 3. Period 3 only applies to those subjects in Part B)
  Plasma PK samples will be collected pre-dose (within 15 minutes prior to dosing) and at 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 36, and 48 hours post- dose.

SECONDARY OUTCOMES:
• Safety and tolerability parameters as assessed by change from baseline in 12-lead ECG and vital signs (BP and HR), number of subjects with adverse events and toxicity grading of clinical laboratory tests. | Up to 28 days
Plasma DTG, ABC and 3TC PK parameters tlag, tmax, t½, Terminal elimination phase rate constant, %AUCex, CL/F and Vz/F, and DTG C24 | For 48 hours after dosing on Day 1 of Periods 1, 2 and 3. Period 3 only applies to those subjects in Part B)
  Plasma PK samples will be collected pre-dose (within 15 minutes prior to dosing) and at 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 36, and 48 hours post- dose.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, Overland Park, Kansas, United States

REFERENCES:
- [Derived] Weller S, Chen S, Borland J, Savina P, Wynne B, Piscitelli SC. Bioequivalence of a dolutegravir, abacavir, and lamivudine fixed-dose combination tablet and the effect of food. J Acquir Immune Defic Syndr. 2014 Aug 1;66(4):393-8. doi: 10.1097/QAI.0000000000000193. PMID 24798770